CLINICAL TRIAL: NCT02177695
Title: A Randomized Phase II Study of Co-Expression Extrapolation (COXEN) With Neoadjuvant Chemotherapy for Localized, Muscle-Invasive Bladder Cancer
Brief Title: S1314, Co-expression Extrapolation (COXEN) Program to Predict Chemotherapy Response in Patients With Bladder Cancer
Acronym: COXEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1314; S1314 (Other: SWOG); NCI-2014-00850 (Other: National Cancer Institute); U10CA180888 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-30 (Estimated); Results first posted 2022-01-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Neoadjuvant Chemotherapy; Coexpression Extrapolation; COXEN; S1314; SWOG
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; Methotrexate; Vinblastine; Doxorubicin; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine & Cisplatin (Experimental): Gemcitabine, 1000 mg/m2, IV, Days 1&8, q 21 days x 4 cycles Cisplatin, 70 mg/m2, IV, Day 1, q 21 days x 4 cycles
  Interventions: Drug: Gemcitabine; Drug: Cisplatin
- Dose Dense MVAC (Experimental): Methotrexate, 30 mg/m2, IV, Day 1, q 14 days x 4 cycles Vinblastine, 3 mg/m2, IV, Day 1 or 2, q 14 days x 4 cycles Doxorubicin, 30 mg/m2, IV, Day 1 or 2, q 14 days x 4 cycles Cisplatin, 70 mg/m2, IV, Day 1 or 2, q 14 days x 4 cycles Filgrastim, 5 mcg/kg, SubQ/IV, Days 3-7, q 14 days x 4 cycles
  Interventions: Drug: Cisplatin; Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Filgrastim

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine, 1000 mg/m2, IV (in the vein) on Days 1 and 8 of each 21 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Gemzar
  Arms: Gemcitabine & Cisplatin
Drug: Cisplatin — Cisplatin, 70 mg/m2, IV (in the vein) on Day 1 of each 21 day cycle (or Day 1 or 2 of each 14 day cycle).
  Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Platinol
Drug: Methotrexate — Methotrexate, 30 mg/m2, IV (in the vein) on Days 1 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Trexall
  Arms: Dose Dense MVAC
Drug: Vinblastine — Vinblastine, 3 mg/m2, IV (in the vein) on Days 1 or 2 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Velban
  Arms: Dose Dense MVAC
Drug: Doxorubicin — Doxorubicin, 30 mg/m2, IV (in the vein) on Days 1 or 2 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Adriamycin
  Arms: Dose Dense MVAC
Drug: Filgrastim — Filgrastim, 5 mcg/kg, SubQ/IV (in the vein) on Days 3-7 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Neupogen
  Arms: Dose Dense MVAC

SUMMARY:
The primary focus of this study is to see if looking at tumor biomarkers using a program called coexpression extrapolation or "COXEN" may predict a patient's response to chemotherapy before surgery.

DETAILED DESCRIPTION:
The COXEN program will not select a patient's therapy, but the type of chemotherapy that he/she will receive will be randomly decided. The patient's response to chemotherapy will be used to test the usefulness of the COXEN program, which is the main goal of this trial. Other potential tests to predict a patient's response to chemotherapy will also be evaluated. In this study, the patient may receive the treatment in Arm 1 (gemcitabine and cisplatin) or the treatment in Arm 2 [methotrexate, vinblastine, doxorubicin, cisplatin, and filgrastim (or pegfilgrastim)]. There will be about 230 people taking part in this study (115 in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven bladder cancer (pure small cell carcinoma, pure adenocarcinoma, and pure squamous cell carcinoma histologies are excluded).
* Stage cT2-T4a N0 M0 disease.
* Documented muscle invasive disease with at least one of the following: disease measuring at least 10 mm on cross-sectional imaging OR the presence of tumor-associated hydronephrosis.
* Staging scans with abdominal/pelvic CT or MRI scan and CT scan or x-ray of the chest within 56 days prior to registration. If alkaline phosphatase is above the treating institution's upper limit of normal (ULN), presence of suspicious bone pain, or if other clinical suspicion, a whole body bone scan is required within 56 days prior to registration.
* Performance status = 0 or 1
* 18 years of age or older
* Must have tumor tissue from transurethral resection of the bladder tumor (TURBT) available for submission that is sufficient for COXEN testing and must agree to submission of 20 (10 micron) slides plus 2 (5 micron) slides from the start and end of the 20 slides for a total of 22 unstained slides.
* Must agree to collection of tissue (if residual disease is present), urine, and whole blood.
* Must agree to participate in the translational medicine studies outlined in the protocol

Exclusion Criteria:

* Prior systemic cytotoxic chemotherapy or systemic anthracycline
* Peripheral neuropathy >/= Grade 2
* Class III/IV heart failure or known left ventricular ejection fraction (LVEF) < 50%
* Clinically relevant hearing impairment > Grade 2
* Renal function, calculated creatinine clearance < 60 mL/min
* Hepatic function, total bilirubin > 1.5 x institutional upper limit of normal (IULN) (or > 2.5 x IULN with Gilbert's disease); AST & ALT > 2 X IULN
* Hematologic function, absolute neutrophil count (ANC) < 1,500/mcL, hemoglobin < 9 g/dL, and platelets < 100,000/mcL
* Hypersensitivity to cisplatin, gemcitabine, doxorubicin, vinblastine, methotrexate, or filgrastim/pegfilgrastim
* Incidence of or uncontrolled medical illness (e.g. active cardiac symptoms, active systemic infection, etc.)
* Pregnant or nursing females
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years. However, patients with localized prostate cancer who are being followed by an active surveillance program are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-08-28 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Flaig, M.D., Study Chair — University of Colorado, Denver
Locations (566):
- United States (566):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Yuma Cancer Center, Yuma, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Stanford Cancer Institute, Palo Alto, California
  - PCR Oncology, Pismo Beach, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Center South Bay, San Jose, California
  - City of Hope South Pasadena, South Pasadena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Cleveland Clinic-Weston, Weston, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Memorial and Saint Elizabeth's Health Care Services LLP, Swansea, Illinois
  - Reid Health, Richmond, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Heartland Cancer Center, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - North Shore Hematology Oncology Associates Inc, Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Maine Center for Cancer Medicine-Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute?Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton Health Center, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Botsford General Hospital, Farmington, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Hematology Oncology Associates East PC, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center - Saint Peters, City of Saint Peters, Missouri
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive
Time Frame: Indefinite
Access Criteria: NCTN/NCORP Data Archive registration
URL: http://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Bai Z, Osman M, Brendel M, Tangen CM, Flaig TW, Thompson IM, Plets M, Scott Lucia M, Theodorescu D, Gustafson D, Daneshmand S, Meeks JJ, Choi W, Dinney CPN, Elemento O, Lerner SP, McConkey DJ, Faltas BM, Wang F. Predicting response to neoadjuvant chemotherapy in muscle-invasive bladder cancer via interpretable multimodal deep learning. NPJ Digit Med. 2025 Mar 22;8(1):174. doi: 10.1038/s41746-025-01560-y. PMID 40121304
- [Derived] Flaig TW, Tangen CM, Daneshmand S, Alva AS, Lucia MS, McConkey DJ, Theodorescu D, Goldkorn A, Milowsky MI, Bangs R, MacVicar GR, Bastos BR, Fowles JS, Gustafson DL, Plets M, Thompson IM Jr, Lerner SP. Long-term Outcomes from a Phase 2 Study of Neoadjuvant Chemotherapy for Muscle-invasive Bladder Cancer (SWOG S1314; NCT02177695). Eur Urol. 2023 Sep;84(3):341-347. doi: 10.1016/j.eururo.2023.06.014. Epub 2023 Jul 4. PMID 37414705
- [Derived] Flaig TW, Tangen CM, Daneshmand S, Alva A, Lerner SP, Lucia MS, McConkey DJ, Theodorescu D, Goldkorn A, Milowsky MI, Bangs R, MacVicar GR, Bastos BR, Fowles JS, Gustafson DL, Plets M, Thompson IM Jr. A Randomized Phase II Study of Coexpression Extrapolation (COXEN) with Neoadjuvant Chemotherapy for Bladder Cancer (SWOG S1314; NCT02177695). Clin Cancer Res. 2021 May 1;27(9):2435-2441. doi: 10.1158/1078-0432.CCR-20-2409. Epub 2021 Feb 10. PMID 33568346

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 237 participants were enrolled, but 10 were ineligible due to missing tissue, inadequate disease assessment and inadequate kidney function.
Groups:
- Gemcitabine & Cisplatin: Gemcitabine, 1000 mg/m2, IV, Days 1&8, q 21 days x 4 cycles Cisplatin, 70 mg/m2, IV, Day 1, q 21 days x 4 cycles
  Gemcitabine: Gemcitabine, 1000 mg/m2, IV (in the vein) on Days 1 and 8 of each 21 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Cisplatin: Cisplatin, 70 mg/m2, IV (in the vein) on Day 1 of each 21 day cycle (or Day 1 or 2 of each 14 day cycle).
  Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
- Dose Dense MVAC: Methotrexate, 30 mg/m2, IV, Day 1, q 14 days x 4 cycles Vinblastine, 3 mg/m2, IV, Day 1 or 2, q 14 days x 4 cycles Doxorubicin, 30 mg/m2, IV, Day 1 or 2, q 14 days x 4 cycles Cisplatin, 70 mg/m2, IV, Day 1 or 2, q 14 days x 4 cycles Filgrastim, 5 mcg/kg, SubQ/IV, Days 3-7, q 14 days x 4 cycles
  Cisplatin: Cisplatin, 70 mg/m2, IV (in the vein) on Day 1 of each 21 day cycle (or Day 1 or 2 of each 14 day cycle).
  Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Methotrexate: Methotrexate, 30 mg/m2, IV (in the vein) on Days 1 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Vinblastine: Vinblastine, 3 mg/m2, IV (in the vein) on Days 1 or 2 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Doxorubicin: Doxorubicin, 30 mg/m2, IV (in the vein) on Days 1 or 2 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Filgrastim: Filgrastim, 5 mcg/kg, SubQ/IV (in the vein) on Days 3-7 of each 14 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
Period: ITT Analysis
Arm/Group | Gemcitabine & Cisplatin | Dose Dense MVAC
Started | 120 | 117
Completed | 115 | 112
Not Completed | 5 | 5
Not completed — Ineligible | 5 | 5
Period: Primary COXEN Analysis
Arm/Group | Gemcitabine & Cisplatin | Dose Dense MVAC
Started | 115 | 112
Participants Excluded From Primary COXEN Analysis | 33 | 27
Completed | 82 | 85
Not Completed | 33 | 27
Not completed — inadequate tissue submitted | 5 | 6
Not completed — insufficient amount of chemotherapy received | 15 | 8
Not completed — Pathologic response not evaluated | 13 | 13

BASELINE CHARACTERISTICS:
Population: All eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine & Cisplatin | Dose Dense MVAC | Total
Number analyzed (Participants) | 115 | 112 | 227
Age, Continuous [Median (Full Range); unit: years] | 64.9 [34.5 to 79.2] | 64.8 [33.1 to 86.5] | 64.8 [33.1 to 86.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 36
  Male | 92 | 99 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 104 | 105 | 209
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 94 | 107 | 201
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 2 | 12
Clinical stage [Count of Participants; unit: Participants] — Clinical T staging based on the TURBT sample and imaging studies
  T2- tumor invades muscularis propia T3- tumor invades perivesical tissue T4a- tumor invades prostatic stroma, uterus, vagina
  Participants
    T2 | 102 | 98 | 200
    T3 or T4a | 13 | 14 | 27
Zubrod performance status [Count of Participants; unit: Participants] — 0- fully active, able to carry out all pre-disease performance without restriction
  1- restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature
  Participants
    0 | 88 | 86 | 174
    1 | 27 | 26 | 53
GC-COXEN score [Count of Participants; unit: Participants] — Coexpression extrapolation (COXEN) score to predict tumor response to treatment with GC.
  COXEN algorithm is a novel approach to generate predictive gene expression models for cancer therapy response. COXEN scores(coefficient) for a participant on a therapy were categorized into low/high scores. High scores predict whether a participant has a 'favorable' response-either pT0 (complete disappearance of tumor) or downgrading to <= pT1 (tumor invades subepithelial connective tissue)- and vice versa for low scores, where 'not favorable' response is having neither a pT0 or <= pT1 predicted response. Population: 47 participants included in the ITT analysis (n=28 on the GC arm, n=19 on the ddMVAC arm) were not evaluable for the primary COXEN analysis and therefore did not have COXEN scores generated
  Participants
    number analyzed (Participants) | 82 | 85 | 167
    Favorable | 18 | 25 | 43
    Not favorable | 64 | 60 | 124
ddMVAC-COXEN score [Count of Participants; unit: Participants] — Coexpression extrapolation (COXEN) score to predict tumor response to treatment with ddmVAC. COXEN algorithm is a novel approach to generate predictive gene expression models for cancer therapy response. COXEN scores(coefficient) for a participant on a therapy were categorized into low/high scores. High scores predict whether a participant has a 'favorable' response-either pT0 (complete disappearance of tumor) or downgrading to <= pT1 (tumor invades subepithelial connective tissue)- & vice versa for low scores, where 'not favorable' response is having neither a pT0 or <=pT1 predicted response. Population: 47 participants included in the ITT analysis (n=28 on the GC arm, n=19 on the ddMVAC arm) were not evaluable for the primary COXEN analysis and therefore did not have COXEN scores generated
  Participants
    number analyzed (Participants) | 82 | 85 | 167
    Favorable | 23 | 30 | 53
    Not Favorable | 59 | 55 | 114

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Whether the Treatment-specific COXEN Score is Prognostic of pT0 Rate
Description: The proportion of participants achieving pT0 in both favorable and unfavorable treatment specific-COXEN score categories.
  Unit of measure is the number of participants in each category that achieved pT0
  _____________________________________________________________________________________________________________________
  The relationship of dose-dense methotrexate, vinblastin, doxorubicin, and cisplatin (DDMVAC)- and gemcitabine+cisplatin (GC)- specific CO-eXpression ExtrapolatioN (COXEN) scores
  This will be done in two ways:
  * By assessing whether the treatment-specific COXEN score is prognostic of pT0 rate or ≤ pT1 in this patient population and to assess in a preliminary fashion whether the COXEN score is a predictive factor distinguishing between these two chemotherapy regimens. .
  * By evaluating the correlation between the GC- and the DDMVAC-COXEN score.
Time Frame: Up to 5 years post registration
Population: Eligible participants that were evaluable for COXEN analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine & Cisplatin | Dose Dense MVAC
Number analyzed (Participants) | 82 | 85
Participants
  Favorable treatment-COXEN score: number analyzed (Participants) | 18 | 30
  Favorable treatment-COXEN score | 8 | 10
  Unfavorable treatment-COXEN score: number analyzed (Participants) | 64 | 55
  Unfavorable treatment-COXEN score | 20 | 17
Statistical Analysis 1: Comparison: Gemcitabine & Cisplatin; To determine the relationship of GC COXEN scores to pT0, GC COXEN score (dichotomous, favorable vs. unfavorable) was tested in a logistic regression model predicting the outcome of pT0 within the GC treatment group; Test type: Superiority; p = 0.1, Regression, Logistic; Odds Ratio (OR) = 2.63, 95% CI 2-sided [0.82 to 8.36]
Statistical Analysis 2: Comparison: Dose Dense MVAC; To determine the relationship of ddMVAC COXEN scores to pT0, ddMVAC COXEN score (dichotomous, favorable vs. unfavorable) was tested in a logistic regression model predicting the outcome of pT0 within the ddMVAC treatment group; Test type: Superiority; p = 0.82, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.42 to 2.95]

2. Primary Outcome: Assessment of Whether the Treatment-specific COXEN Score is Prognostic of ≤ pT1 Rate
Description: The proportion of participants achieving <=pT1 in both favorable and unfavorable treatment specific-COXEN score categories.
  Unit of measure is the number of participants in each category that achieved <= pT1
  ____________________________________________________________________________________________________________________ The relationship of dose-dense methotrexate, vinblastin, doxorubicin, and cisplatin (DDMVAC)- and gemcitabine+cisplatin (GC)- specific CO-eXpression ExtrapolatioN (COXEN) scores
  This will be done in two ways:
  * By assessing whether the treatment-specific COXEN score is prognostic of pT0 rate or ≤ pT1 in this patient population and to assess in a preliminary fashion whether the COXEN score is a predictive factor distinguishing between these two chemotherapy regimens. .
  * By evaluating the correlation between the GC- and the DDMVAC-COXEN score.
Time Frame: up to 5 years post-registration
Population: Eligible participants that were evaluable for COXEN analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine & Cisplatin | Dose Dense MVAC
Number analyzed (Participants) | 82 | 85
Participants
  Favorable treatment-COXEN score: number analyzed (Participants) | 18 | 30
  Favorable treatment-COXEN score | 10 | 16
  Unfavorable treatment-COXEN score: number analyzed (Participants) | 64 | 55
  Unfavorable treatment-COXEN score | 30 | 31
Statistical Analysis 1: Comparison: Gemcitabine & Cisplatin; To determine the relationship of GC COXEN scores to <= pT1, GC COXEN score (dichotomous, favorable vs. unfavorable) was tested in a logistic regression model predicting the outcome of pT1 or better within the GC treatment group; Test type: Superiority; p = 0.02, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.11 to 4.89]
Statistical Analysis 2: Comparison: Dose Dense MVAC; To determine the relationship of ddMVAC COXEN scores to <=pT1, ddMVAC COXEN score (dichotomous, favorable vs. unfavorable) was tested in a logistic regression model predicting the outcome of pT1 or better within the ddMVAC treatment group; Test type: Superiority; p = 0.76, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.46 to 1.75]

3. Primary Outcome: Assessment of COXEN Score as a Predictive Factor Distinguishing Between GC and ddMVAC
Description: To assess in a hypothesis generating fashion, the ability of COXEN to select for an individual chemotherapy regimen (GC vs DDMVAC)
  P-values are reported as a measure of whether COXEN can select between GC/DDMVAC and to determine the significance of interactions between treatment specific COXEN scores and treatment arms in models predicting either pT0 or <= pT1. Interactions with p-values > 0.05 are interpreted as not significant.
  ________ The relationship of dose-dense methotrexate, vinblastin, doxorubicin, and cisplatin (DDMVAC)- and gemcitabine+cisplatin (GC)- specific CO-eXpression ExtrapolatioN (COXEN) scores
  This will be done in two ways:
  * By assessing whether the treatment-specific COXEN score is prognostic of pT0 rate or ≤ pT1 in this patient population and to assess in a preliminary fashion whether the COXEN score is a predictive factor distinguishing between these two chemotherapy regimens. .
  * By evaluating the correlation between the GC- and the DDMVAC-COXEN score.
Time Frame: up to 5 years post-registration
Population: Eligible participants that were evaluable for COXEN analysis. Participants in this arm were pooled to test the ability of the COXEN algorithm to distinguish between GC and ddMVAC treatment, with the assumption that there is no interaction between the COXEN score and treatment arm.
Measure: Number; unit: p-value
Groups:
- All Participants: Eligible participants that were evaluable for COXEN analysis
Arm/Group | All Participants
Number analyzed (Participants) | 167
p-value
  P-value of interaction term (GCscore*treatment arm) in model predicting pT0 | 0.88
  P-value of interaction term (GCscore*treatment arm) in logistic regression model predicting <=pT1 | 0.43
  P-value of interaction term (MVACscore*treatment arm) in logistic regression model predicting pT0 | 0.66
  P-value of interaction term (MVACscore*treatment arm) in logistic regression model predicting <=pT1 | 0.85

4. Primary Outcome: Correlation Between GC-and ddMVAC-COXEN Score
Description: The Pearson and Spearman correlation coefficients for GC-and ddMVAC-COXEN score were calculated and are reported below.
  ___________________________________________________________________________________________________________________ The relationship of dose-dense methotrexate, vinblastin, doxorubicin, and cisplatin (DDMVAC)- and gemcitabine+cisplatin (GC)- specific CO-eXpression ExtrapolatioN (COXEN) scores
  This will be done in two ways:
  * By assessing whether the treatment-specific COXEN score is prognostic of pT0 rate or ≤ pT1 in this patient population and to assess in a preliminary fashion whether the COXEN score is a predictive factor distinguishing between these two chemotherapy regimens. .
  * By evaluating the correlation between the GC- and the DDMVAC-COXEN score.
Time Frame: up to 5 years post-registration
Population: as for outcome 3
Measure: Number; unit: correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 167
correlation coefficient
  Pearson correlation coefficient | 0.385
  Spearman correlation coefficient | 0.386

5. Secondary Outcome: Predictability of the CO-eXpression ExtrapolatioN (COXEN) Score to Direct Which of the Two Regimens the Patient Should Receive: Gemcitabine+Cisplatin (GC) Versus Dose-dense Methotrexate, Vinblastin, Doxorubicin, and Cisplatin (DDMVAC)
Description: In addition to stratification factors and dichotomous COXEN GEM score, an indicator for treatment arm and the interaction of treatment arm with COXEN GEM score was also included in a logistic regression model. A significant interaction would suggest that the respective COXEN GEM score was able to differentiate whether a patient was more likely to respond to one chemotherapy regimen over another. *note that this is the same objective at Primary Outcome #3 above - this was erroneously listed twice in the protocol.
Time Frame: Up to 5 years post registration
Population: as for outcome 3
Measure: Number; unit: p-value
Arm/Group | All Participants
Number analyzed (Participants) | 167
p-value
  Pvalue of interaction term (GCscore*treatment arm) in model predicting pT0 | 0.88
  Pvalue of interaction term (GCscore*treatment arm) in model predicting <=pT1 | 0.43
  Pvalue of interaction term (MVACscore*treatment arm) in model predicting pT0 | 0.66
  Pvalue of interaction term (MVACscore*treatment arm) in model predicting <=pT1 | 0.85

6. Secondary Outcome: Value of Gene Expression Profiling in Predicting Overall Survival (OS)
Description: 5-year OS curve was estimated using the Kaplan-Meier method. Included all COXEN evaluable participants regardless of arm assignment. The report groups were favorable vs. unfavorable COXEN status.
Time Frame: Up to 5 years post registration
Population: Eligible participants across both arms that were evaluable for COXEN analysis.
Measure: Number; unit: Percent of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 167
Percent of Participants
  Favorable COXEN Status: number analyzed (Participants) | 48
  Favorable COXEN Status | 76
  Unfavorable COXEN Status: number analyzed (Participants) | 119
  Unfavorable COXEN Status | 71

7. Secondary Outcome: Pathologic T0 Rate Evaluation: Gemcitabine+Cisplatin (GC) Versus Dose-dense Methotrexate, Vinblastin, Doxorubicin, and Cisplatin (DDMVAC)
Description: Pathologic complete response rate at the time of cystectomy following GC or DDMVAC treatment
Time Frame: Up to 5 years post-registration
Population: Participants who received treatment in Gemcitabine & Cisplatin and Dose Dense MVAC arms.
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine & Cisplatin | Dose Dense MVAC
Number analyzed (Participants) | 82 | 85
percentage of participants | 36 | 42

8. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported. Grade 3 is less severe than Grade 5.
  Grade 3 - Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL* (bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden).
  Grade 4 - Life-threatening consequences; urgent intervention indicated. Grade 5 - Death related to AE
  *ADL- Activities of Daily Living
Time Frame: Duration of treatment and follow up until death or 5 years post registration
Population: Participants who received at least one dose of protocol treatment, submitted toxicity data and were included in the ITT analysis.
Measure: Number; unit: Participants
Groups:
- Gemcitabine and Cisplatin: Gemcitabine, 1000 mg/m2, IV, Days 1 and 8, q 21 days x 4 cycles Cisplatin, 70 mg/m2, IV, Day 1, q 21 days x 4 cycles
  Gemcitabine: Gemcitabine, 1000 mg/m2, IV (in the vein) on Days 1 and 8 of each 21 day cycle. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Cisplatin: Cisplatin, 70 mg/m2, IV (in the vein) on Day 1 of each 21 day cycle (or Day 1 or 2 of each 14 day cycle).
  Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
Arm/Group | Gemcitabine and Cisplatin | Dose Dense MVAC
Number analyzed (Participants) | 115 | 112
Participants
  Acute kidney injury | 0 | 1
  Alanine aminotransferase increased | 1 | 0
  Anemia | 10 | 9
  Bronchial infection | 0 | 1
  Cardiac arrest | 0 | 1
  Cardiac disorders - Other, specify | 1 | 0
  Chronic kidney disease | 2 | 1
  Creatinine increased | 0 | 5
  Dehydration | 0 | 2
  Diarrhea | 0 | 2
  Dizziness | 1 | 0
  Dyspnea | 1 | 0
  Enterocolitis infectious | 0 | 1
  Erectile dysfunction | 1 | 0
  Esophagitis | 0 | 1
  Fall | 0 | 1
  Fatigue | 3 | 5
  Febrile neutropenia | 2 | 2
  Headache | 0 | 1
  Heart failure | 0 | 1
  Hematuria | 0 | 1
  Hyperglycemia | 3 | 2
  Hyperkalemia | 2 | 0
  Hypertension | 1 | 3
  Hypocalcemia | 0 | 1
  Hypokalemia | 0 | 3
  Hypomagnesemia | 0 | 2
  Hyponatremia | 5 | 2
  Hypophosphatemia | 1 | 0
  Infections and infestations - Other, specify | 0 | 3
  Insomnia | 0 | 1
  Investigations - Other, specify | 0 | 1
  Kidney infection | 1 | 0
  Lung infection | 0 | 1
  Lymphocyte count decreased | 2 | 3
  Mucositis oral | 0 | 5
  Nausea | 1 | 3
  Neutrophil count decreased | 20 | 10
  Phlebitis infective | 1 | 0
  Platelet count decreased | 11 | 5
  Proteinuria | 1 | 0
  Renal and urinary disorders - Other, specify | 1 | 0
  Sepsis | 0 | 1
  Syncope | 1 | 1
  Thromboembolic event | 4 | 1
  Tinnitus | 1 | 0
  Upper gastrointestinal hemorrhage | 0 | 1
  Urinary tract infection | 4 | 3
  Urinary tract obstruction | 1 | 1
  Vestibular disorder | 0 | 1
  Vomiting | 0 | 3
  White blood cell decreased | 5 | 6

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post registration
Description: Participants who received protocol treatment and are included in the ITT analysis
Arm/Group | Gemcitabine and Cisplatin | Dose Dense MVAC
All-Cause Mortality (participants affected / at risk) | 28/115 | 25/112
Serious Adverse Events (participants affected / at risk) | 1/115 | 4/112
Other Adverse Events (participants affected / at risk) | 112/115 | 108/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Cisplatin (N=115) | Dose Dense MVAC (N=112)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Sudden death NOS (General disorders) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Cisplatin (N=115) | Dose Dense MVAC (N=112)
Anemia (Blood and lymphatic system disorders) | 83 | 69
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac disorders-Other (Cardiac disorders) | 1 | 2
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Heart failure (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 9 | 3
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 1 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 4 | 7
Tinnitus (Ear and labyrinth disorders) | 18 | 25
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 6 | 6
Conjunctivitis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Eye disorders-Other (Eye disorders) | 0 | 2
Photophobia (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 12 | 10
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Anal pain (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 47 | 46
Diarrhea (Gastrointestinal disorders) | 19 | 27
Dry mouth (Gastrointestinal disorders) | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 10
Dysphagia (Gastrointestinal disorders) | 2 | 2
Esophageal pain (Gastrointestinal disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 11 | 16
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 4 | 4
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 12 | 39
Nausea (Gastrointestinal disorders) | 65 | 72
Oral dysesthesia (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 1 | 4
Stomach pain (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 18 | 28
Chills (General disorders) | 4 | 4
Edema face (General disorders) | 0 | 2
Edema limbs (General disorders) | 16 | 13
Fatigue (General disorders) | 82 | 77
Fever (General disorders) | 12 | 5
Flu like symptoms (General disorders) | 5 | 1
General disorders and admin site conditions - Other (General disorders) | 4 | 4
Infusion related reaction (General disorders) | 1 | 1
Infusion site extravasation (General disorders) | 1 | 0
Injection site reaction (General disorders) | 4 | 1
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 1
Malaise (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 4 | 3
Pain (General disorders) | 7 | 8
Allergic reaction (Immune system disorders) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 2
Eye infection (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 2 | 5
Kidney infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Phlebitis infective (Infections and infestations) | 2 | 0
Rash pustular (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 2 | 3
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 17 | 11
Bruising (Injury, poisoning and procedural complications) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 10 | 8
Alkaline phosphatase increased (Investigations) | 16 | 23
Aspartate aminotransferase increased (Investigations) | 6 | 7
Blood bilirubin increased (Investigations) | 0 | 1
Cholesterol high (Investigations) | 0 | 2
Creatinine increased (Investigations) | 34 | 37
Hemoglobin increased (Investigations) | 1 | 1
Investigations-Other (Investigations) | 4 | 3
Lymphocyte count decreased (Investigations) | 18 | 16
Neutrophil count decreased (Investigations) | 44 | 15
Platelet count decreased (Investigations) | 50 | 37
Weight gain (Investigations) | 5 | 0
Weight loss (Investigations) | 11 | 11
White blood cell decreased (Investigations) | 42 | 14
Anorexia (Metabolism and nutrition disorders) | 28 | 35
Dehydration (Metabolism and nutrition disorders) | 10 | 9
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 25 | 29
Hyperkalemia (Metabolism and nutrition disorders) | 10 | 10
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 | 24
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 11 | 20
Hypomagnesemia (Metabolism and nutrition disorders) | 35 | 38
Hyponatremia (Metabolism and nutrition disorders) | 25 | 29
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 7
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 3
Obesity (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 11 | 9
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Concentration impairment (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 15 | 17
Dysgeusia (Nervous system disorders) | 19 | 24
Headache (Nervous system disorders) | 18 | 19
Memory impairment (Nervous system disorders) | 1 | 2
Nervous system disorders-Other (Nervous system disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 1 | 3
Peripheral motor neuropathy (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 14
Presyncope (Nervous system disorders) | 2 | 0
Sinus pain (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 3 | 4
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 3 | 2
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 13 | 3
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 23 | 16
Libido decreased (Psychiatric disorders) | 1 | 0
Psychiatric disorders-Other (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 7
Bladder spasm (Renal and urinary disorders) | 2 | 2
Chronic kidney disease (Renal and urinary disorders) | 6 | 3
Cystitis noninfective (Renal and urinary disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 17 | 13
Proteinuria (Renal and urinary disorders) | 4 | 2
Renal and urinary disorders-Other (Renal and urinary disorders) | 4 | 3
Urinary frequency (Renal and urinary disorders) | 14 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 2
Urinary tract pain (Renal and urinary disorders) | 7 | 8
Urinary urgency (Renal and urinary disorders) | 2 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 3 | 3
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Hiccups (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 48
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 6
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 7
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Social circumstances-Other (Social circumstances) | 1 | 2
Flushing (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 2 | 3
Hypertension (Vascular disorders) | 23 | 30
Hypotension (Vascular disorders) | 5 | 2
Phlebitis (Vascular disorders) | 2 | 0
Superficial thrombophlebitis (Vascular disorders) | 2 | 0
Thromboembolic event (Vascular disorders) | 11 | 4
Vascular disorders-Other (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02177695/Prot_SAP_ICF_000.pdf